CLINICAL TRIAL: NCT02095756
Title: A Randomized, Split-Face, Double-Blind Clinical Pilot Study of Combination Picosecond Alexandrite Laser and Non-Hydroquinone Topical Therapy Versus Topical Therapy Alone for the Treatment of Facial Melasma
Brief Title: Combination Alexandrite Laser and Topical Therapy vs Topical Therapy Alone for Treatment of Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PICO-2013-01
Record Dates: First submitted 2014-03-17; First posted 2014-03-26 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 755nm Alexandrite laser (Experimental): 755nm Alexandrite laser for the treatment of melasma
  Interventions: Other: 755nm Alexandrite Laser and Lytera Skin Brightening System (Non-Hydroquinone Topical Therapy); Other: Lytera Skin Brightening System (Non-hydroquinone topical therapy)

INTERVENTIONS:
Other: 755nm Alexandrite Laser and Lytera Skin Brightening System (Non-Hydroquinone Topical Therapy)
Other: Lytera Skin Brightening System (Non-hydroquinone topical therapy)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a combination of non-hydroquinone topical therapy and a 755nm Alexandrite compared to topical therapy alone for the treatment of facial melasma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Subjects aged 18-74 years of age;
* Fitzpatrick Skin Types I-IV;
* Female subjects of childbearing potential must have a negative urine pregnancy test at the beginning of the study, and agree to practice appropriate birth-control to prevent pregnancy during the study. The type and dose of birth control must have been stable for at least 3 months prior to study entry and it is not expected to change during the study; acceptable methods of birth control are oral contraceptives, contraceptive patches/rings/implants Norplant®, Depo-Provera®, double-barrier methods (e.g. condoms and spermicide), abstinence and vasectomies of partner with a documented second acceptable method of birth control should the subject become sexually active.
* Subjects diagnosed with moderate to severe melasma on both sides of the face
* For subjects using medication to treat a concurrent medical condition, type and dose must have been stable for at least 3 months prior to study entry and it is not expected to change during the study (except any medications specifically outlined in the exclusion criteria section)
* Subjects able to avoid prolonged sun exposure on the face for the duration of the study and willing to use appropriate sun avoidance techniques.
* Subjects able to follow study instructions and likely to complete all required visits;
* Subjects/Representative able and willing to sign the Informed Consent (which includes a photography release) prior to any study procedures.

Exclusion Criteria:

* Female subjects who are pregnant, nursing or planning a pregnancy during the course of the study;
* Subjects with a condition or who are in a situation which, in the Investigator's opinion, may put the Subject at risk, may confound the study results, or may interfere with the Subject's participation in the study, such as: the use of a concomitant medication that can interfere with the study or worsen any condition when used during the study, the use of medications known to induce photosensitivity;
* Subjects under treatment for a dermatologic condition, which may interfere with the safe evaluation of the study regimen (e.g. eczema, psoriasis, severe sun-damage, dermatitis) and/or have scarring or infection of the area to be treated;
* Subjects with a diagnosis of skin cancer (BCE, SCC, Melanoma, etc.) in the areas to be treated;
* Subject unwilling to avoid any other treatment for melasma during the study (total duration of 30 weeks);
* Subjects with a wash-out period of less than 14 days for melasma treatments at the time of study entry or under current treatment;
* Subjects with prior facial resurfacing, deep or chemical peels within 6 months of the date of study entry;
* Subject unwilling to refrain from any facial cosmetic procedures during the study period (e.g., chemical peels, resurfacing, microdermabrasion, etc.);
* Subject has initiated treatment with hormones including estrogen, progesterone and/or oral contraceptives within 3 months of study entry, or who intend to discontinue hormonal therapy during the study;
* Subject has participated in a clinical research study within the last 30 days prior to enrollment;
* Subject is unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or other reasons;
* Subject is unable to meet the study attendance requirements.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Melasma clearance | up to 3 months post last treatment
  Evaluate the efficacy of a combination of non-hydroquinone topical therapy and a 755-nm alexandrite laser compared to topical therapy alone in the treatment of melasma .

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc., San Diego, California, United States